CLINICAL TRIAL: NCT04695236
Title: A Prospective, Multicenter, Randomized Clinical Trial to Evaluate the Safety and Efficacy of Intravascular Hypothermia Therapy of Patients With Acute Ischemic Stroke
Brief Title: A Trial of Intravascular Hypothermia Therapy in Acute Ischemic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: jiaoliqun (Other)
Responsible Party: Sponsor-Investigator, jiaoliqun, Prof., Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASPIRE
Record Dates: First submitted 2021-01-01; First posted 2021-01-05 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Hypothermia; Reperfusion Injury; Ischemic Stroke; Thrombectomy
MeSH Terms: conditions — Hypothermia; Reperfusion Injury; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessment by independent investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Study Group: Intravascular hypothermia therapy group ZOLL Intravascular Temperature Management system, Quattro catheter will be used in study group
  Interventions: Device: ZOLL Intravascular Temperature Management system, Quattro catheter
- Control group (Placebo Comparator): Control group: Without intravascular hypothermia therapy group
  ZOLL Intravascular Temperature Management system, Quattro catheter will not be used in control group
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Device: ZOLL Intravascular Temperature Management system, Quattro catheter — ZOLL Intravascular Temperature Management system, Quattro catheter
  Arms: Study group
Other: Standard Treatment — Standard Treatment for Ischemic Strokre
  Arms: Control group

SUMMARY:
Acute ischemic stroke (AIS) has been one of the major causes of global mortality and morbidity. The superiority of endovascular therapy (EVT) over standard medical therapy in treating AIS due to large vessel occlusion (LVO) in the anterior circulation has been widely accepted. However, a critical concern is that even with an extremely high rate of successful recanalization (the modified thrombolysis in cerebral infarction [mTICI] score 2b-3) around 90%, nearly half of the patients failed to benefit from EVT. So, adjunctive therapy of EVT for neuroprotection is required.

From the previous domestic and foreign literatures, hypothermia can prevent and treat secondary injury caused by ischemia-reperfusion injury and cerebral edema of acute cerebral ischemia, so as to achieve the role of neuroprotection. In this study, intravascular cooling was performed as soon as possible with careful temperature control in patients receiving thrombectomy. The temperature was controlled at 33° C for 48-72 hours. This parallel controlled study is to systematically evaluate the feasibility and safety of adjunctive therapy using early intravascular hypothermia in AIS patients receiving mechanical thrombectomy. The results will clarify a potential modality for neuroprotection and hopefully provide new evidence in improving patient prognosis.

DETAILED DESCRIPTION:
In this study, the target subjects were AIS patients with successful recanalization (mTICI 2b-3). Early intravascular hypothermia neuroprotection therapy was given to patients after thrombectomy to evaluate its safety and effectiveness. The neuroprotection effect of endovascular hypothermia therapy is explored regarding several aspects, such as hemorrhagic conversion rate, cerebral edema, and neurological function recovery, with specific evaluation criteria described in detail in the following experimental design.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old
2. Clinical signs consistent with acute ischemic stroke with large vessel occlusion in the anterior circulation (internal carotid artery, middle cerebral artery M1 or M2 segment)
3. ASPECTS score 0-10
4. Arterial puncture could be performed within 24 hours from symptom onset or LKN
5. Baseline NIHSS (NIHSS) score prior to randomization ≥ 10 and NIHSS 1a ≥ 1
6. Candidate for endovascular thrombectomy therapy in accordance with best practices per AHA standard stroke guidelines meeting all labeling requirements for EVT in the trial
7. Successful recanalization of occluded vessel (mTICI 2b-3) after EVT
8. No intracranial hemorrhage postoperative CT examinations immediately after recanalization. If the subject' recanalization of vessel could not achieve mTICI 2b-3, the subject could not enter the per-protocol analysis and will separate another group
9. Informed consent form signed by subjects or their legal guardian

Exclusion Criteria:

1. Subject who suffer serious infection (e.g. sepsis) or multiple organ failure
2. Known presence of an IVC filter
3. End stage renal disease on hemodialysis
4. Known hypersensitivity to antiplatelet agents, anticoagulation drugs, iodinated contrast and/or anesthetics
5. Known hypersensitivity to the components of the medical device
6. Any known history of the following conditions: bleeding diathesis, coagulopathy, cryoglobulinemia, sickle cell anemia, will refuse blood transfusions or contraindication to heparin; history of genetically confirmed hypercoagulable syndrome
7. Use of warfarin with INR > 3
8. Hemodynamically significant cardiac dysrhythmias (eg. QTc interval >450 msec, bradycardia (heart rate less than 50), Mobitz Type II second degree AV block (or higher AV block), and severe ventricular dysrhythmias (sustained VT or VF)) which cause significant hypotension (SBP ≤ 120 mmHg requiring more than two pressor medications)
9. Platelet count<40×10^9/L
10. Blood glucose concentration <2.7 or > 22.2 mmol/L
11. Hypertension uncontrollable by drug treatment (systolic blood pressure≥185 mmHg or diastolic blood pressure≥110mmhg)
12. Expected life expectancy<6 months
13. Temperature < 35°C on admission to Emergency Department
14. With a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations (e.g., dementia or mental illness)
15. Subject participating in a study involving an investigational drug or device that would impact the current study
16. Baseline CT/MR evidence of multiple vascular territory acute stroke
17. Baseline CT/MR showing evidence of arterial vasculitis or dissection
18. Evidence of intracranial hemorrhage or hemorrhagic transformation before thrombectomy
19. Evidence of intracranial hemorrhage or hemorrhagic transformation immediately after thrombectomy
20. Presence of pulmonary embolism, ilio-femoral or deep vein thrombosis
21. Brain vascular lesion (e.g. aneurysm or arteriovenous malformation)
22. Brain tumor or CNS infection
23. Concurrent participation in a study involving an investigational drug or device that would impact the current study
24. Female patient of childbearing potential who is known to be pregnant or lactating
25. For other reasons, the researchers believe that the patient is not suitable for continued treatment
26. Patients without a legally authorized representative to sign the consent form will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Intracranial hemorrhage conversion rate | 7 days after thrombectomy operation or discharge
  ICH

SECONDARY OUTCOMES:
Modified Rankin scale (mRS) | 90 days
  The mRS is a 7-point scale ranging from 0 (no symptoms) to 6 (death)
The rate of functional independency (mRS 0-2) | 90 days
  The mRS is a 7-point scale ranging from 0 (no symptoms) to 6 (death)
The rate of mortality (mRS 6) | 90 days
  The mRS is a 7-point scale ranging from 0 (no symptoms) to 6 (death)
NIHSS | 24 hours, 7 days or discharge
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits.
Rate of symptomatic intracranial hemorrhage (sICH) | 7 days after thrombectomy operation or discharge
  The diagnosis of sICH was based on the association of ICH with any of the following. conditions: (1) Increase in NIHSS score > 4 points compared to the score before ICH; (2) Increase in NIHSS score by >2 points in one category; (3) deterioration leading to intubation, hemicraniectomy, external ventricular drain placement, or any other major interventions.
Rate of malignant cerebral edema | 7 days after thrombectomy operation or discharge
  Development of signs of herniation (including decrease in consciousness and/or anisocoria), accompanied by midline shift >= 5 mm on follow-up imaging.
Infarct volume | 5-7 days after thrombectomy operation or discharge
  measured on 5-7 days CT (or MRI if available)

OTHER OUTCOMES:
Rate of any major adverse events | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao,MD, PhD, Principal Investigator — Department of Neurosurgery & Interventional Neuroradiology Xuanwu Hospital
Locations (1):
- Xuanwu Hospital, Beijing, China